CLINICAL TRIAL: NCT03491007
Title: Neurosteroids in PTSD - Biomarkers to Therapeutics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI obtained outside employment that was not compatible with this award
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-021-17S; 1IK2CX001397-01A2 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; DHEA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, double-blind, placebo (PBO)-controlled, randomized Phase 2 pilot study using adjunctive dehydroxyepiandrosterone [DHEA (400 mg)] will be evaluated to establish Proof of Concept (POC) for this agent in Veterans with PTSD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo (PBO)-controlled, randomized Phase 2 pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (No Intervention): Subjects will receive a one-time oral dose of PBO prior to initial brain imaging followed by sustained administration of PBO for 6 weeks.
- DHEA (Placebo Comparator): Subjects will receive a one-time oral dose of DHEA prior to initial brain imaging followed by sustained administration of DHEA for 6 weeks.
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA — Subjects will be randomized to receive a one-time oral dose of DHEA (400mg) or PBO and sustained administration of the study drug for 6 weeks. There will be a 2 week placebo lead-in period [all participants], followed by subjects continuing in the randomization block of DHEA or placebo for 6 weeks following acute administration).
  Arms: DHEA

SUMMARY:
The purpose of this research is to determine if a study medication called Dehydroepiandrosterone (DHEA) helps to reduce PTSD symptoms in OEF/OIF/OND Veterans. In addition to finding out if DHEA is effective for treating PTSD symptoms, this research seeks to determine if DHEA is effective in treating other symptoms, such as depression and anxiety. Depression and anxiety are symptoms that are frequently present in Veterans who are experiencing PTSD. Another purpose of this research is to takes pictures of the brain using magnetic resonance imaging (MRI) and blood levels of various small molecules including neurosteroids and also proteins, which may be affected by the study drug and/or related to symptoms in Veterans with PTSD. This study seeks to determine if DHEA is changed to other compounds after it is taken by mouth and the safety and effectiveness of DHEA in Veterans with PTSD. This is an "add-on" study and Veterans enrolled in the study will continue to take all of their current medications without any changes (also called "usual care"), and DHEA or a sugar pill (also called a "placebo") will then be added to their current medication regimen.

DETAILED DESCRIPTION:
This is a parallel-group, double-blind, placebo (PBO)-controlled, randomized Phase 2 pilot study using adjunctive dehydroxyepiandrosterone [DHEA (400 mg)] to establish Proof of Concept (POC) for use of this agent in Veterans with PTSD.

The investigators' first objective is POC target engagement to evaluate a one-time adjunctive oral dose of DHEA (400 mg) relative to PBO on the neuronal circuity of fear-anxiety-emotion connectivity. This will be achieved by comparing pre- to post-treatment changes in amygdala-hippocampal functional connectivity to DHEA and PBO during fMRI activation. The investigators hypothesize that compared with PBO, DHEA will increase task-associated fMRI functional connectivity between the amygdala and hippocampus (primary outcome).

The second objective is to determine if an 8-week treatment with adjunctive DHEA is superior to PBO in reducing symptoms of PTSD (CAPS-5) and depression (BDI) in OEF/OIF/OND Veterans, and enhancing resilience (CD-RISC). The investigators hypothesize that 400mg DHEA will result in reduced PTSD and depression symptom severity relative to PBO, as determined by a pre- to post-treatment decrease in CAPS-5 and BDI scores, respectively, with enhancement in resilience scores using the CD-RISC at 6-weeks.

The third objective is to evaluate the impact of DHEA relative to PBO on serum neurosteroid levels in OEF/OIF/OND Veterans with PTSD. The investigators hypothesize that DHEA will result in a statistically-significant increase in serum neurosteroid levels (DHEA, DHEAS, androsterone) relative to PBO, as determined by pre- to post-treatment reductions in PTSD symptoms severity. This association will be evaluated by correlating neurosteroid levels with PTSD, depression, and resilience scores over 6 weeks of treatment.

The exploratory objective is to determine preliminary evidence for an association of fMRI and myelin integrity measures of fear-anxiety-emotion circuits with serum neurosteroid levels and treatment response to DHEA. Changes in myelin integrity following DHEA treatment will be evaluated using novel susceptibility diffusion imaging [STI]), as DHEA impacts myelination in preclinical rodent models. The investigators will also determine if serum neurosteroid levels are correlated with myelin integrity on STI. The investigators hypothesize that fMRI and myelin integrity of fear-anxiety circuits will correlate with serum neurosteroids and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND era Veterans
* PTSD diagnosis (CAPS-5 score 33).
* Negative pregnancy test if female.

  * Sexually active subjects are required to use a medically acceptable form of birth control if they are of childbearing potential and could become pregnant during the study.
  * A medically acceptable form of birth control includes non-hormonal intrauterine devices, surgical sterilization, or double barrier methods (e.g., diaphragm with contraceptive jelly, condom with contraceptive foam, cervical caps with contraceptive jelly).
  * Sexual abstinence with agreement to continue abstinence or to use a medically acceptable method of contraception should sexual activity occur is permissible.
* Female participants must have had a normal mammogram within the last year (if older than 40)
* Female participants must have had a normal pelvic exam within the last year
* No change in medications less than 4 weeks before baseline assessment
* No anticipated need to alter medications for PTSD for the 6-week study duration (as determined by study physician's review of records and/or discussion with prescribing physician).
* Ability to fully participate in the informed consent process

Exclusion Criteria:

* Unstable medical or neurological illness, including seizures, renal impairment or CVA and inability to participate in neuroimaging (fMRI).
* Use of oral contraceptives or other hormonal supplements, as it is unclear if DHEA metabolism to other neurosteroids such as estradiol may potentially impact contraceptive efficacy.
* Significant suicidal or homicidal ideation.
* Current DSM-5 diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder (including major depression with psychotic features), or cognitive disorder due to a general medical condition.
* Female patients who are pregnant or breast-feeding.
* Known allergy to study medication.
* History of moderate or severe TBI.
* Substance dependence within past three months, per DSM-5 criteria (excluding caffeine and nicotine).
* Abnormal prostate specific antigen (PSA; >2.5ng/ml in males age 49 or less; >4ng/ml in males age 50 or greater) or history of prostate cancer, breast cancer, or uterine cancer.
* A family history of prostate, breast or endometrial cancer in a first-degree relative.
* Presence of any factors/conditions, medical or non-medical, that may interfere with conduction of study assessments in the judgment of the study team.
* Serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions or behaviors that would compromise participation and/or likely to lead to worsening of symptoms during the course of the study in the opinion of study physician and research team.
* Are non-ambulatory or require the use of crutches or a walker.
* Taking Narcotic medications or benzodiazepines for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Szabo, MD PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DHEA
Started | 3 | 2
Completed | 0 | 1
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DHEA | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.33 (2.87) | 34.00 (5) | 34.2 (3.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity Between Amygdala-hippocampus Assessed Using fMRI Based Shifted-attention Emotion Appraisal (SEAT) Paradigm.
Description: The Shifted-Attention Emotion Appraisal (SEAT) Paradigm will present compound stimuli that include both emotional faces (e.g. sad, happy, angry) and neutral scenes. In three different conditions, participants are asked to respond to three different questions: (1) 'Gender'; (2) 'Inside/Outside'; or (3) 'Like/Dislike'. This allows multiple components of cognition to be probed including (1) implicit emotional processing, (2) attentional modulation, and (3) cognitive modulation of emotion. Item-specific memory will be tested first using yes/no recognition judgments. The conjunctive memory test will require participants to make "match" (previously viewed faces and buildings presented in a combinations seen during encoding) or "mismatch" (items in combinations not previously seen together) judgments. Change in SEAT paradigm (Z score) from baseline to 6 weeks
Time Frame: 6 weeks
Population: Neuroimaging data not available. Software setup and code creation for fMRI analyses was intended to occur after all participants had been enrolled and all scans had been performed (and available to be analyzed). Study was terminated prior to full participation and the data needed was simply not collected.
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to make a diagnosis of PTSD and assess PTSD symptoms. It assesses the intensity and frequency of PTSD symptoms. Change in total CAPS-5 score from baseline to 6 weeks. Scores range from 0-80; higher score indicates greater severity.
Time Frame: Baseline and 6 weeks
Population: Study was terminated prior to analysis (PI obtained outside employment that was not compatible with this award).
  Only one participant completed the study (randomized to DHEA); only this one participant thus had data for the primary outcome measure (change from baseline to study completion for primary endpoint).
  Only one other participant had post-randomization data (randomized to placebo x 2 weeks then withdrew from study).
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -5

3. Secondary Outcome: Beck-Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item self-report inventory of depression symptoms. The minimum and maximum values for the BDI-II are (0-63). Change in total BDI-II score from baseline to 6 weeks. Higher score indicates greater severity.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -12

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The HAM-A is clinician-rated interview that measures presence of anxiety-related symptoms in 14 areas. Total score ranges from 0 to 56. Higher score indicates greater anxiety. Change in total HAM-A score from baseline to 6 weeks
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -3

5. Secondary Outcome: Symptom Checklist-90-Revised (SCL-90-R)
Description: Change in total SCL-90-R score (range: 90 to 450; higher score indicates greater severity) from baseline to 6 weeks. This scale assesses somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -8

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity Scale
Description: PROMIS Pain Intensity is a three item scale measuring the severity of pain using a five-point Likert-type scale (i.e., no pain=1, mild=2, moderate=3, severe=4, very severe=5).Change in total PROMIS Pain Intensity Scale score (range: 3 to 15) from baseline to 6 weeks. Higher score indicates greater severity.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | 0

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Scale
Description: The 8-item PROMIS Sleep Disturbance measures sleep disturbance with each item on the measure rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8-40. Change in total PROMIS-Sleep Disturbance score from baseline to 6 weeks. Higher score indicates greater severity.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | 1

8. Secondary Outcome: PROMIS-Anger Scale
Description: The PROMIS-Anger Scale is an 8-item scale that assesses anger. Scores range from 5 to 25, with higher scores indicating greater anger severity. Change in total PROMIS-Anger score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | 0

9. Secondary Outcome: Barrat Impulsivity Scale (BIS-11)
Description: The BIS-11 is a 30 item questionnaire to measure impulsiveness. Items are answered on a 4-point scale. Total scores range from 30-120 with a higher summed score indicating higher impulsivity. Change in total BIS-11 score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -15

10. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: The CD-RISC scale assesses resiliency in individuals. There are 25 items in the survey, each item is scored from 0-4, and the total ranges from 0-100. Higher scores indicate greater resilience. Change in total CD-RISC score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | 20

11. Secondary Outcome: Hamilton Depression Ratings Scale (HAM-D)
Description: The HAM-D is a standardized, clinician-administered rating scale; assesses 17 items characteristically associated with major depression. Total scores range from 0-50. Higher score indicates greater severity. Change in total HAM-D score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | 2

12. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression Scale
Description: PROMIS-Depression Scale is a self-reported scale of depressive symptoms Each item is scored 1-5 (1 = Never; 5 = Always). Total ranges are 8 to 40. Higher score indicates greater severity. Change in total PROMIS Depression score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -2

13. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety Scale
Description: The PROMIS-Anxiety Scale is a self-report of anxiety symptoms. Each item is scored 1-5 (1 = Never; 5 = Always). Total score ranges from 8 to 40. Higher score indicates greater severity. Change in total PROMIS Anxiety score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -4

14. Secondary Outcome: Clinician Global Impression Scale (CGI)
Description: The CGI scale will be used to rate improvement in the subject's condition. Total score range of 0-30. Higher scores indicates greater severity. Change in total CGI score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -3

15. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) assesses the severity of pain and its impact on functioning. Total range of 0-110. Higher score indicates greater severity. Change in total BPI score from baseline to 6 weeks.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: score on a scale (change score)
Arm/Group | Placebo | DHEA
Number analyzed (Participants) | 0 | 1
score on a scale (change score) |  | -5

16. Other Pre Specified Outcome: Serum DHEA
Description: Change in serum levels of DHEA from baseline to 6 weeks
Time Frame: 6 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Myelin Integrity Susceptibility Tensor Imaging (STI)
Description: Change in STI (Z score) from baseline to 6 weeks
Time Frame: 6 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Serum DHEAS
Description: Change in serum DHEAS levels from baseline to 6 weeks
Time Frame: 6 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Serum Androsterone
Description: Change in serum androsterone levels from baseline to 6 weeks
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected at each visit throughout study participation and by phone two weeks post study completion, up to 10 weeks.
Arm/Group | Placebo | DHEA
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | DHEA (N=2)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Restlessness (General disorders) | 1 (1) | 0 (0)
Decreased Appetite (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03491007/Prot_SAP_000.pdf